CLINICAL TRIAL: NCT06200389
Title: Epidemiological Study of Vulvovaginal Candidiases Strain Types and Risk Factors Among Gynecological Outpatients From Multiple Sites in China
Brief Title: Epidemiological Study of Vulvovaginal Candidiases Strain Types and Risk Factors Among Gynecological Outpatients in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MA-VVC-EI-001
Record Dates: First submitted 2023-12-28; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-10

CONDITIONS: Vulvovaginal Candidiases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fungal culture and drug sensitivity detection of vaginal secretions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: microbiology testing — Vulvovaginal Candidiases patients diagnosed by microbiology testing can be included

SUMMARY:
We has proposed to conduct a national epidemiological study on the pathogenic strains and high risk factors of Vulvovaginal Candidiasis in China , and conduct drug resistance analysis.

DETAILED DESCRIPTION:
Vulvovaginal Candidiasis is a mucosal infectious disease, which rarely occurs fatal infection, but has high recurrence rate. Vulvovaginal Candidiasis often leads to decreased life quality and serious economic burden. However, we known little about the pathogenesis of Vulvovaginal Candidiasis. So better diagnosis and treatment methods are needed to decrease the impact on women's health.

In 2017, the national Vulvovaginal Candidiasis epidemiological survey led by Professor Liao showed that 543 strains of fungi were isolated from different patients from 12 hospitals in 10 cities in China, of which Recurrence Vulvovaginal Candidiasis strains accounted for 15.7%. The most common pathogenic strain was Candida albicans (460 species, 84.71%), and the most common non-albicans was Candida glabra (47 species, 8.66%). In addition, 92 isolates (20.4%) belonged to the new branch endemic to North China. Vaginal symptoms of Vulvovaginal Candidiasis caused by non-albicans are usually milder compared to Vulvovaginal Candidiasis caused by Candida albicans. However, inherent resistance to azoles, as well as acquired resistance mechanisms, can complicate the treatment of non-albicans and often requires a long-term antifungal treatment or other treatments to clear non-albicans.

Given that the resistance rate of different types of candida to antifungal drugs changes over time, common antifungal drugs have selective induction of resistance to fungi, and fungi have cross-induction of resistance to antifungal drugs, it is very important to evaluate the distribution and resistance of Candida species in a long-term . Accurate and effective acquisition of candida epidemiological data to understand the recent status and drug resistance of Candida infection can effectively guide clinical treatment to improve the therapy, and play a very important role in clinical diagnosis and treatment. Therefore, Professor Liao has proposed to conduct a national epidemiological study on the pathogenic strains and high risk factors of Vulvovaginal Candidiasis in China once again, and conduct drug resistance analysis, in order to guide clinicians to better Vulvovaginal Candidiasis treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients of gynecology
2. Age≧18 years
3. Signed informed consent form voluntarily
4. With diagnosis and symptomatology of Vulvovaginal Candidiasis (all types of Vulvovaginal Candidiasis can be included)
5. History of sexual life

Exclusion Criteria:

1. Antifungal medication was used within 7 days (oral or topical)
2. With contraindications of vaginal sampling
3. Other conditions deemed unsuitable for inclusion by clinicians

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with Vulvovaginal Candidiasis symptomatology and positive culture
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Composition and distribution of strains from gynecological Vulvovaginal Candidiasis outpatients in China | From January 2024 to January 2025

SECONDARY OUTCOMES:
Evaluate the sensitivity and resistance of commonly used antifungal treatments | From January 2024 to January 2025
Evaluate risk factors of gynecological Vulvovaginal Candidiasis outpatients in China | From January 2024 to January 2025
Estimate the proportion of different ages of gynecological Vulvovaginal Candidiasis outpatients in China (Childbearing age and non-childbearing age) | From January 2024 to January 2025
Consistency analysis of clinical and microbiological diagnosis from gynecological Vulvovaginal Candidiasis outpatients in China | From January 2024 to January 2025
Estimate the proportion of various types of Vulvovaginal Candidiasis in gynecological outpatients in China | From January 2024 to January 2025
Evaluate neuropsychic behaviour of Vulvovaginal Candidiasis patients in gynecological outpatients nationwide | From January 2024 to January 2025